CLINICAL TRIAL: NCT02584374
Title: Balloon Test for Iliac Vein Compression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL54330
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-10

CONDITIONS: May-thurner Syndrome
Keywords: iliac vein compression
MeSH Terms: conditions — May-Thurner Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: with suspected iliac vein compression, but with no signs of compression on venography and if venography with balloon occlusion test is performed.
  Interventions: Other: Venography with balloon occlusion test
- Healthy controls: Healthy subjects between 18-45 years of age
  Venography with balloon occlusion test will be performed.
  Interventions: Other: Venography with balloon occlusion test

INTERVENTIONS:
Other: Venography with balloon occlusion test — First, regular venography of the venous iliac tract will be performed. Second, a 16mm diameter balloon will be inflated in the common iliac vein and venography will be repeated.

SUMMARY:
Iliac vein compression is a common cause of leg or abdominal complaints and is difficult to diagnose. Although a combination of duplex ultrasonography, magnetic resonance venography and two-plane phlebography are able to show compression, not all suspected iliac vein compressions can be identified. Intravascular ultrasound appears to have a higher diagnostic value, but is far more expensive. In our experience a balloon occlusion test in the common iliac vein during phlebography can diagnose iliac vein compression due to the collateral network that is visualised. The general consensus is that pelvic collaterals are a sign of pathology, though the investigators would like to validate this test by showing that a balloon occlusion test in healthy subjects does not identify a collateral network.

DETAILED DESCRIPTION:
Rationale: Iliac vein compression is a common cause of leg or abdominal complaints and is difficult to diagnose. Although a combination of duplex ultrasonography, magnetic resonance venography and two-plane phlebography are able to show compression, not all suspected iliac vein compressions can be identified. Intravascular ultrasound appears to have a higher diagnostic value, but is far more expensive. In the investigators' experience a balloon occlusion test in the common iliac vein during phlebography can diagnose iliac vein compression due to the collateral network that is visualised. The general consensus is that pelvic collaterals are a sign of pathology, though the investigators would like to validate this test by showing that a balloon occlusion test in healthy subjects does not identify a collateral network.

Objective: The objective of this study is to identify whether venography with balloon occlusion of the common iliac vein has value in the diagnosis of iliac vein compression syndrome.

Study design: This is an observational study in healthy subjects compared to a patient population with suspected iliac vein compression.

Study population: Healthy subjects between the ages of 18 and 45 and patients with suspected iliac vein compression who show no signs of compression on venography.

Diagnostic test: Subjects will undergo a diagnostic phlebography, during which the common iliac vein is occluded by balloon inflation and contrast is injected to identify whether a network of pelvic collaterals will appear.

Main study parameters/endpoints: The main endpoint of this study is the presence of collaterals that cross the midline after balloon occlusion of the left common iliac vein, which is scored as present or not Additionally, a quantitive analysis of collaterals will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (all patients who have been diagnosed using this technique will be used as a comparison group)

Exclusion Criteria:

* Disease affecting the circulatory system, such as cardiac disease, varicosities or peripheral arterial disease, on the basis of anamnesis.
* History of bleeding or clotting disorders
* Complaints of the abdomen or leg consistent with iliac vein compression syndrome or pelvic congestion syndrome
* Clinical-Etiologic-Anatomic-Pathophysiologic classification of C2 or higher (C0: no venous signs, C1: venectasia, C2: varicose veins, C3: edema, C4: skin changes, C5 healed ulcer, C6: active ulcer)
* History of deep venous thrombosis or pulmonary embolism.
* History of surgery of the abdomen, groin or lower limb
* Pregnancy
* Allergy to contrast or lidocaine
* Active malignancy
* (For the patient comparison group: obvious signs of compression on venography without balloon occlusion test)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers (all patients who have been diagnosed using this technique will be used as a comparison group)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Presence of collaterals (prevalence number) | During venography
  During regular venography the presence and amount of collaterals are scored. Collaterals need to cross the midline to be considered positive. Subsequently, balloon occlusion of the left common iliac vein will be performed and another contrast injection will take place. The presence and amount of collaterals will again be assessed. Quantitive analysis will be performed to evaluate the amount of collaterals and how they are branched off.

CONTACTS AND LOCATIONS:
Overall Officials: R de Graaf, MD, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Netherlands